CLINICAL TRIAL: NCT05271435
Title: Digital Tools for Assessment of Motor Functions and Falls in ALS
Status: Active, not recruiting | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: BioSensics (Industry)
Responsible Party: Principal Investigator, Andrew Geronimo, Assistant Research Professor, Dept of Neurosurgery, Milton S. Hershey Medical Center
Other Study IDs: STUDY13892
Record Dates: First submitted 2022-01-12; First posted 2022-03-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-01

CONDITIONS: ALS; PLS; PMA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: PAMSys Activity Monitoring System — This system is composed of a Study Tablet running custom fall detection and reporting software and PAMSys sensors. PAMSys provides clinical-grade physical activity monitoring, storing the raw accelerometer data that can be used for analyzing activity parameters such as those listed in Table 3. Sensor data will be downloaded manually upon receipt of the study device by Biosensics, the study sponsor. Sensors can be worn during all activities including while showering and sleeping. The rated battery life is 3-6 months for the fall sensor, and 4 weeks for the activity sensors. This system is not classified as a medical device. Reports of sensor use, step number, battery level, and memory availability are sent hourly to a secured and HIPAA compliant back-end server provided by BioSensics. The Study Tablet also contains modules for performing speech, handwriting, and pattern tracing tasks.
Behavioral: Motor, Speech, and Handwriting Assessment — These assessments occur at each study visit. After equipping the subject with 3 activity sensors (1 on pendant around neck and 2 on wrists).
  * 10-meter walk task (5 minutes) - The subject starts from a standing position and walks a length of 10 meters. The best time of three trials is used.
  * Timed Up and Go (TUG) test (5 minutes) - Subjects stand, walk to a marker on the floor 3 meters ahead, turn around the marker, walk back to the chair, and sit. The best time of three trials is used.
  * Handwriting Assessment Battery (HAB) (15 minutes) [Faddy2008] - The subject is seated at a table with a pencil and paper and performs a series of writing tasks.
  * Speech Assessment Battery (SAB)(10 minutes) - The participant will perform a set of audio recordings using the study tablet while sitting in a quiet room.

SUMMARY:
This is a 48-week single arm study that incorporates digital tools for assessing motor function as part of an ALS telemonitoring program. During the study, neck- and wrist-worn "activity sensors" (PAMSys, BioSensics, Newton, MA) that will be worn by subjects while performing tasks of daily living. Subjects will also complete a motor, speech, and handwriting assessment during site visits. Subjects will complete a digital home assessments of speech, handwriting, and pattern tracing tasks throughout the study, and report any falls which occur on the study tablet. The investigators will explore whether functional changes are sensitive to self-reported changes on the ALS Functional Rating Scale - Revised (ALFRS-R) over the length of the study.

DETAILED DESCRIPTION:
Many of the recognized intrinsic factors for falls are commonly seen in ALS, including advanced age, muscle weakness, gait and balance problems, and previous falls. The American Academy of Neurology ALS Quality Standards Committee recommends querying patients for falls occurring in the past 12 months, indicating that prevention of falls is an important part of disease management. Despite this, the determinants and prevention of falls in this population is critically understudied.

Among frail older adults, fallers (those who reported at least 1 fall in the last 6-months) spent more than twice as much time walking as non-fallers (those who reported no falls in the last 6-months). For these individuals, the best predictors of falling are measures related to activity exposure, such as time spent walking, average walking bout duration, or steps per day. Activity metrics of cadence variability, peak vertical acceleration variability, average duration of episodes of walking, frontal acceleration variability, average peak vertical acceleration, and average cadence have been shown to be associated with fall risk. During walking, individuals with ALS have increased and highly variable gait cycle time (time to complete a full walking cycle), along with reduced stride length with increased variability in stride length compared to healthy controls.

The ability to observe changes in gait and posture has rapidly advanced around a revolution in mobile health technology. Inertial measurement units (IMUs), a standard inclusion of nearly all new smartphone/smartwatch devices, are small electronic chips that detect different aspects of inertial change, notably linear acceleration, angular velocity, and position relative to the magnetic field of the earth. Unlike their expansive use in movement disorders like Parkinson's disease, IMU-based gait assessment has been largely absent in ALS, despite the rapid changes to gait that may occur. The standard model for assessing and acting upon functional motor changes, including those impacting gait and falls, occurs roughly once every three months when patients are seen in the outpatient setting. Furthermore, self-reporting of falls has been shown to suffer from recall bias, resulting in low sensitivity and underreporting of fall events. In summary, patients with a rapidly progressing neurodegenerative disease, who in the standard care setting receive physical assessment motor function every three months, might stand to benefit from a home-based, objective biomarker for functional motor changes.

ELIGIBILITY:
Inclusion Criteria

1. Diagnosis of definite, probable, probable laboratory-supported, or possible ALS by revised El Escorial research criteria [Brooks2000], primary lateral sclerosis (PLS), or progressive muscular atrophy (PMA).
2. 18 years of age or older;
3. ALSFRS-R walking sub-score of either 4 (normal gait), 3 (early ambulation difficulties), or 2 (walking with assistance);
4. Fluent in written and spoken English.

Exclusion Criteria

1. Neurological or orthopedic problems independent of their inclusionary diagnosis that affects their gait;
2. Pregnant or nursing woman;
3. Prisoner or institutionalized individuals;
4. Have any clinically relevant medical history of other disease or diseases that, in the opinion of the research team, exclude the subject from participation (including severe cognitive dysfunction).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with motor neuron disease experiences changes in their walking.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Physical Activity at 10 months | baseline and visit 4 (an average of 10 months)
  Changes in physical activity from baseline to 10 months will be assessed. Physical activity will be quantified by measuring number of taken steps per day and will be measured using a validated wearable sensor named PAMSys. Monitoring of physical activity will be done during 72 hours at baseline and 72 hours at 10 months.

SECONDARY OUTCOMES:
Change from baseline in total lower limb muscle strength at end of study | baseline and end of study (an average of 1 year)
  Strength testing is performed by the attending neurologist at clinical appointments. Bilateral hip flexion, knee extension and flexion, and foot dorsiflexion strength will be documented according to Medical Research Council (MRC) grade 0 (no power) to 5 (normal power). Total score for bilateral muscle groups ranges from 0 to 40. Change in total lower limb strength score over study period will be calculated.
Change from baseline in total upper limb muscle strength at end of study | baseline and end of study (an average of 1 year)
  Strength testing is performed by the attending neurologist at clinical appointments. Bilateral deltoids, biceps, triceps, wrist extension, and interossei strength will be documented according to Medical Research Council (MRC) grade 0 (no power) to 5 (normal power). Total score for bilateral muscle groups ranges from 0 to 50. Change in total upper limb strength score over study period will be calculated.
Change from baseline in total upper limb reflexes at end of study | baseline and end of study (an average of 1 year)
  Reflex testing is performed by the attending neurologist at clinical appointments. Bilateral biceps, triceps, and brachioradialis reflexes will be documented according to Modified Ashworth Scale grade 0 (no tone increase) to 4 (limb rigid). Total score for bilateral muscle groups ranges from 0 to 24. Change in total upper limb reflexes over study period will be calculated.
Change from baseline in total lower limb reflexes at end of study | baseline and end of study (an average of 1 year)
  Reflex testing is performed by the attending neurologist at clinical appointments. Bilateral patellar and achilles reflexes will be documented according to Modified Ashworth Scale grade 0 (no tone increase) to 4 (limb rigid). Total score for bilateral muscle groups ranges from 0 to 16. Change in total lower limb reflexes over study period will be calculated.
Change from baseline in Forced Vital Capacity at end of study | baseline and end of study (an average of 1 year)
  Forced vital capacity (FVC) is collected at clinical appointments. FVC is expressed as a percentage (%) of predicted volume against an age, height, and ethnicity matched standard. Change in FVC over this time period will be calculated.
Change from baseline in total ALSFRS-R at end of study | baseline and end of study (an average of 1 year)
  ALS Functional Rating Scale-Revised (ALSFRS-R) measures function in 12 domains. The total score ranges from 48 (normal function) to 0 (no function). Change in total score over this time period will be calculated.
Change from baseline in ALSFRS-R gross motor subscore at end of study | baseline and end of study (an average of 1 year)
  ALS Functional Rating Scale-Revised (ALSFRS-R) gross motor subscore measures function in 3 domains. The total subscore ranges from 12 (normal function) to 0 (no function). Change in total subscore over this time period will be calculated.
Change from baseline in ALSFRS-R fine motor subscore at end of study | baseline and end of study (an average of 1 year)
  ALS Functional Rating Scale-Revised (ALSFRS-R) fine motor subscore measures function in 3 domains. The total subscore ranges from 12 (normal function) to 0 (no function). Change in total subscore over this time period will be calculated.
Change from baseline in "Falls Efficacy Scale - International" total score at end of study | baseline and end of study (an average of 1 year)
  The Falls Efficacy Scale - International (FES-I) is collected at study visits. The total score ranges from 64 (high concern about falling) to 0 (no concern about falling). Change in total score over this time period will be calculated.
Change from baseline in "Fatigue Severity Scale" total score at end of study | baseline and end of study (an average of 1 year)
  The Fatigue Severity Scale is collected at study visits. The total score ranges from 63 (high fatigue) to 9 (low fatigue). Change in total score over this time period will be calculated.
Change from baseline in "Neurological Fatigue Index - Motor Neuron Disease" weakness subscale at end of study | baseline and end of study (an average of 1 year)
  The Neurological Fatigue Index - Motor Neuron Disease is collected at study visits. The weakness subscale total score ranges from 21 (high fatigue) to 7 (low fatigue). Change in total score over this time period will be calculated.
Change from baseline in "Neurological Fatigue Index - Motor Neuron Disease" energy subscale at end of study | baseline and end of study (an average of 1 year)
  The Neurological Fatigue Index - Motor Neuron Disease is collected at study visits. The energy subscale total score ranges from 18 (high fatigue) to 6 (low fatigue). Change in total score over this time period will be calculated.
Change from baseline in speaking rate at end of study | baseline and end of study (an average of 1 year)
  Subjects will complete the audio recording of a standard reading passage every two weeks. The speaking rate will be calculated from this audio, and the change in speaking rate over the study period will be calculated.
Change from baseline in 3-meter Timed-Up-and-Go at end of study | baseline and end of study (an average of 1 year)
  3-meter timed-up-and-go task is recorded at study visits. The best time of three trials is recorded. Change in best time over the study period will be calculated.
Change from baseline in 10 meter walk at end of study | baseline and end of study (an average of 1 year)
  A 10-meter walk task is recorded at study visits. The best time of three trials is recorded. Change in best time over the study period will be calculated.
Handwriting Assessment: Change from baseline in handwriting speed at end of study | baseline and end of study (an average of 1 year)
  As part of the Handwriting Assessment Battery completed at study visits, subjects will copy a standard sentence from a prompt in the booklet. The change in writing speed for this copying task over the study period will be calculated.
Handwriting Assessment: Change from baseline in legibility at end of study | baseline and end of study (an average of 1 year)
  As part of the Handwriting Assessment Battery (HAB) completed at study visits, subjects will print the alphabet in upper and lowercase, as well as the numbers 1-12. Legibility will be determined as the percent of individual characters rated as legible according to the HAB handbook. The change in character legibility over the study period will be calculated.
Digital Handwriting Assessment: Change from baseline in handwriting speed at end of study | baseline and end of study (an average of 1 year)
  As part of the Digital Handwriting Assessment performed every two weeks on the study tablet, subjects will copy a standard sentence from a prompt on the tablet. The change in writing speed for this copying task over the study period will be calculated.
Digital Handwriting Assessment: Change from baseline in legibility at end of study | baseline and end of study (an average of 1 year)
  As part of the Digital Handwriting Assessment performed every two weeks on the study tablet, subjects will print the alphabet in upper and lowercase, as well as the numbers 1-12. Legibility will be determined as the percent of individual characters rated as legible according to the HAB handbook. The change in character legibility over the study period will be calculated.
Digital Handwriting Assessment: Change from baseline in spiral tracing speed at end of study | baseline and end of study (an average of 1 year)
  As part of the Digital Handwriting Assessment performed every two weeks on the study tablet, subjects will be timed as they trace the outline of a spiral. The change in time to complete the tracing over the study period will be calculated.
Fall Event Detections | end of study (an average of 1 year)
  Fall events (falls and near-falls) detected by the sensor are registered on the study tablet. The total number of fall events registered over the course of the study is a secondary outcome.
Fall Event Reports | end of study (an average of 1 year)
  Subjects enter fall event reports in the study tablet. The total number of reports reported over the course of the study is a secondary outcome
Adherence: Tablet Assessments | end of study (an average of 1 year)
  Total number of assessments (handwriting, speech, and pattern tracing) completed on the tablet over the study period.
Adherence: Fall Sensor | end of study (an average of 1 year)
  Total number of hours registered with wearing the fall sensor over the study period.
Adherence: Activity Sensor | end of study (an average of 1 year)
  Total number of hours registered with wearing the activity sensors over the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No